CLINICAL TRIAL: NCT06909292
Title: A Post-market, Multicenter, Prospective, Clinical Study to Evaluate the Nevro1 Sacroiliac (SI) Transfixing and Fusion System for the Treatment of Sacroiliac Joint Dysfunction
Brief Title: Sacroiliac (SI) Joint Transfixing and Fusion: Meaningful Long Term Outcomes With Nevro1
Acronym: SIMON1
Status: Recruiting | Type: Observational
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: CA2024-02 US SIJ-PM
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Sacroiliac transfixing; sacroiliac fusion; sacroiliac joint pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treated Group: Treated with Nevro1 transfixing and fusion system
  Interventions: Device: Sacroiliac Joint transfixing and fusion system (Nevro1)

INTERVENTIONS:
Device: Sacroiliac Joint transfixing and fusion system (Nevro1) — The Nevro1 is a titanium cage the is implanted in the sacroiliac join from a posterior direction, and then anchors are deployed that stabilize the joint. It has multiple openings to allow surgeons to fill them with autogenous bone graft to encourage bone bridging through the implant for SIJ fusion.

SUMMARY:
The goal of this observational study is to learn if Nevro1 Sacroiliac Transfixing and Fusion System can treat sacroiliac joint dysfunction in males or females over 21. The main questions it aims to answer is what percentage of patients have clinically important pain relief with no adverse events, and what proportion of patients have fusion of the sacroiliac joint at 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Has medical insurance that covers this standard of care procedure and all other anticipated and unanticipated procedure-related care, and all coverage criteria required by insurer are met, which may include but are not limited to:

   * Has had low back and/or buttock pain for at least 6 months that is inadequately responsive to non-surgical care
   * Has a positive Fortin's test
   * Has a diagnosis of SIJ dysfunction (degenerative sacroiliitis or SI disruption) with pain elicited on at least 3 of 5 provocative tests (FABER, Gaenslen, Distraction, Thigh Thrust, Compression).
   * At least 75% reduction in pain for the expected duration of two anesthetics (on separate visits each with a different duration of action), and the ability to perform previously painful maneuvers, following an image-guided, contrast-enhanced intra-articular (diagnostic) SIJ injection
   * A trial of at least one therapeutic intra-articular SIJ injection (i.e. corticosteroid injection)
2. Has an ODI score ≥30% at enrollment
3. Has a SI joint pain score of at least 5 out of 10 on numerical rating scale at enrollment.
4. Be at least 21 years of age at enrollment
5. The patient's physician has decided that the best treatment for the patient's SIJ dysfunction is the Nevro1 SI Fixation System, and the patient has agreed to the treatment
6. Be willing and capable of giving written informed consent
7. Be mentally and physically able to comply with study-related requirements and procedures and attend all scheduled visits

Exclusion Criteria:

1. Has current severe back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, lumbar radicular pain, and lumbar vertebral body fracture
2. Has SIJ pain secondary to inflammatory conditions or other known sacroiliac pathology such as: Sacral dysplasia, inflammatory sacroiliitis (e.g., ankylosing spondylitis or other HLA-associated spondylo-arthropathy), tumor, infection, acute fracture, and crystal arthropathy
3. Has had a previous SIJ implant placement, including an allograft
4. Has had an injection with corticosteroid into the index SIJ within the last 30 days
5. Has had a sacral radiofrequency ablation within the last 6 months
6. Has a history of recent (<1 year) major trauma to pelvis
7. Has previously diagnosed or suspected severe osteoporosis (defined as prior T-score < -2.5 or history of osteoporotic fracture)
8. Has a chronic rheumatologic condition (e.g., rheumatoid arthritis)
9. Has a known allergy to titanium or titanium alloys
10. Has a current local or systemic infection that raises the risk of surgery
11. Is currently receiving or seeking short- or long-term worker's compensation related to the SI joint or low back pain, is currently receiving disability remuneration related to SI joint or low back pain, and/or is currently involved in injury litigation related to the SI joint or low back pain
12. Is participating in an investigational study or has been involved in an investigational study within 3 months prior to enrollment
13. Has any condition or anatomy that makes treatment with the Nevro1 SI Fixation System infeasible
14. Is taking a medication known to have detrimental effects on bone quality and soft tissue healing
15. Has a prominent neurologic condition that would interfere with physical therapy
16. Be pregnant or plan on becoming pregnant in the next two years.
17. Has a medical condition or pain in other area(s), not intended to be treated in this study, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort will be selected from participating clinics
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-04-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Composite Pain Relief and Safety Responder | 6 months
  The proportion of patient meeting the following criteria:
  * NRS score for SIJ pain reduced by at least 2 points from baseline.
  * Absence of implant-related serious adverse events (SAEs).
  * Absence of neurologic worsening related to the lumbosacral nerve roots.
  * Absence of reoperation (removal, revision reoperation or supplemental fixation) for SIJ pain.

SECONDARY OUTCOMES:
Change in Disability | 6 months
  Absolute change from baseline in Oswestry Disability Index (ODI) score. The total score ranges from 0 (minimal disability) to 100 (severe disability, e.g., bedridden).
Patient Global Impression of Change (PGIC) | 6 months
  Proportion of patients reporting "Better" or "A great deal better" on the PGIC. The PGIC is a 7-point scale with responses ranging from "no change (or condition has gotten worse)" to "a great deal better".
Physical and Mental Health Summary (PROMIS-29) | 6 months
  Absolute change from baseline in PROMIS-29 score. Higher scores represent greater impact of pain on a patients life in the domains of physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance.
Change in Quality of Life | 6 months
  Absolute change from baseline in the index score of EuroQol 5-dimension 5 level (EQ-5D-5L) a standardized measure of health status. The index score ranges from zero to one, with one representing the highest possible health state.
Change in Sleep Disturbance Due to Pain | 6 months
  Absolute change from baseline in Pain and Sleep Questionnaire Three-Item Index (PSQ-3) score. The scale ranges from 0 (pain does not affect sleep) to 30 (pain has maximum effect on sleep).
Timed "Up and Go" Performance test (TUG) | 6 months
  Absolute change from baseline in time to perform the TUG.

OTHER OUTCOMES:
Presence of bone apposition on implant surface | 12 and 24 months
  Grading of the presence of bone apposition on the device adjacent to the sacrum and ilium.
Presence of bony fusion across the sacroiliac joint | 12 and 24 months
  Grading of the presence of bony fusion across the sacroiliac joint.
Presence of radiolucency at the implant surface | 12 and 24 months
  Grading of the presence of radiolucency at the device surface adjacent to the sacrum and ilium.
Proportion of patients with different levels of treatment response | 3, 6, 12, and 24 months
  Evaluating different pain relief response rates, defining responder as a participant who experiences ≥30%, ≥50% and ≥80% pain relief vs. Baseline as measured by NRS.
Sub-analysis comparing outcomes between age groups | 3, 6, 12, and 24 months.
  All outcomes will be compared between the two age groups: 21 to 70 years, and 71 years and above.
Rate of adverse events | Implant, 1, 3, 6, 12, and 24 months.
  Proportion of patients who experience and adverse event related to the procedure or device including infection, device breakage, migration, neurological worsening, and procedural blood loss.

CONTACTS AND LOCATIONS:
Overall Officials: Rose P Azalde, MS, Study Director — Nevro Corp
Locations (5):
- United States (5):
  - AIRS Clinic, Lodi, California
  - Michigan Orthopaedic Surgeons, Southfield, Michigan
  - Carolinas Pain Institute, Winston-Salem, North Carolina
  - Advanced Spine and Pain Specialists, Spring, Texas
  - Procura Pain and Spine, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No
Study data will be reported with descriptive statistics describing group level outcomes, not individual outcomes.